CLINICAL TRIAL: NCT01888692
Title: A Prospective Observational Study to Evaluate the Impact of PET/CT Simulation on Radiation Treatment Planning in Relation to Changes in GTV in Locally Advanced Non-small Cell Lung Cancer
Brief Title: To Evaluate the Impact of PET/CT on Radiation Treatment Planning in Relation to Changes in GTV in Stage 3 NSCLC
Status: Terminated | Type: Observational
Why Stopped: Poor accural
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: B2006;089
Record Dates: First submitted 2013-06-18; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
Keywords: PET/CT; Radiotherapy; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Acknowledging that level I evidence already exists regarding the general beneficial impact on FDG PET in the staging and subsequent management of lung cancer the investigators postulate that fusing PET/CT data sets with RT CT simulation data sets for adult patients with conventionally/clinically assessed stage III non-small cell lung cancer will have a significant impact on GTV as well as normal tissue irradiation. This research will also estimate inter and intra-observer variability of treatment planning, relative to GTV, between and amongst radiation oncologists.

DETAILED DESCRIPTION:
Primary objectives of the study:

1.To determine the impact of PET/CT fusion on gross tumor volume ( GTV ) for primary(GTVP) and nodal (GTVN) disease for each patient by comparing GTV contours using two separate data sets.

(A) GTVP CT+ ve and GTVN CT+ ve

(B) GTVP PET+ve and GTVN PET +ve

GTV will be measured and recorded in cubic centimeters for each volume.

Secondary Endpoints:

1.Normal tissue toxicity:3D conformal Computerized radiation plans will be generated for the data sets GTVP and GTVN A and B .Dose Volume Histogram (DVH) will be determined and compared for the following normal tissue toxicity parameters.

I. V 20 Both lungs (Combined total lung volumes including PTV): Volume of both lungs receiving ≥ 20 G y, including planning target volume.

II. Mean lung dose: Mean radiation dose received by both lungs in a given radiation plan, calculated by the planning computer.

III. V 55 Esophagus: Volume of esophagus receiving≥ 55Gy.

IV. Mean esophageal dose : Mean radiation dose received by whole esophagus in a given radiation plan, calculated by the planning computer

V. Spinal cord dose: Maximum dose received by the spinal cord in a given radiation plan.

V1.. V40 Whole heart: Volume of heart receiving ≥ 40Gy

2A Inter observer variation: This will be determined for the data sets GTV A and B only delineated by 4 radiation oncologists blinded to each other, for first 20 patients. The resident involved in this project will be responsible to co-ordinate this part of the project. GTV will be measured and recorded in cubic centimeters for each volume.

2B Intra observer variation: This will be determined for the data sets GTV A and B only delineated by the same radiation oncologist (treating physician) at two different occasions, for first 20 patients. Minimum time interval between the two contours will be one month .The resident involved in this project will be responsible to co-ordinate this part of the project. GTV will be measured and recorded in cubic centimeters for each volume.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be eligible for the Oncology FDG PET Winnipeg PET Program/Edmonton Cross Cancer Institute Extended Phase III Clinical Trial - Protocol 001, and in addition;
* Pathologically proven NSCLC
* Clinical stage III A (inoperable) or stage IIIB where there is intent to pursue radical curative RT/chemo, staged with conventional imaging as outlined in standard work up section.
* ECOG Performance status 0-2
* Age ≥ 18 years
* FEV1 ≥ 1.0 L
* No prior or concurrent malignancy except non-melanomatous skin cancer unless disease-free for one year or more for non primary bronchogenic cancers and two years for primary bronchogencic cancers;
* No prior RT to thorax.
* Must be able to start RT within 4 weeks after PET/CT simulation
* Participants may be treated with radical radiation only or without concurrent chemotherapy, adjuvant chemotherapy or neo-adjuvant therapy.

Exclusion Criteria:

* As per Oncology FDG PET Winnipeg PET Program/Edmonton Cross Cancer Institute Extended Phase III Clinical Trial - Protocol 001 and more specifically:
* Unable/unwilling to give informed consent.
* Uncontrolled hyperglycemia ( Blood sugar> 12 mmol/L)
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically proven NSCLC Clinical stage III A (inoperable) or stage IIIB where there is intent to pursue radical curative RT/chemo, staged with conventional imaging as outlined in standard work up section
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2007-04; Primary Completion 2009-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Impact of PET/CT fusion on gross tumor volume for primary and nodal disease for each patient by comparing GTV contours using three separate data sets. | From April 2007 -upto two years

CONTACTS AND LOCATIONS:
Overall Officials: Naseer Ahmed, MD, Study Director — CancerCare Manitoba
Locations (1):
- Cancer Care Manitoba, Winnipeg, Manitoba, Canada